CLINICAL TRIAL: NCT06498570
Title: Clinical Outcomes of Two Symmetrical Kera-rings Implantation in Grade Three Keratoconus; A Retrospective Non-Randomized Study
Brief Title: Clinical Outcomes of Two Symmetrical Kera-rings Implantation in Grade Three Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Assistant Professor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-MED-24-05--03PD
Record Dates: First submitted 2024-06-28; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Cornea Ectasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- grade 3 keratoconic eyes Grade 3 eyes with stable keratoconus (Other): grade 3 keratoconic eyes Grade 3 eyes with stable keratoconus
  Interventions: Device: Intracorneal rings

INTERVENTIONS:
Device: Intracorneal rings — The (ICRS), intracorneal rings segments implantation surgery
  Other Names: INTACS

SUMMARY:
Clinical Outcomes of Two Symmetrical Kera-rings Implantation in Grade Three Keratoconus

DETAILED DESCRIPTION:
a retrospective non- randomized controlled clinical study. The study included twenty-three grade 3 keratoconic eyes of twenty-three patients, the keratoconus staging was based on Amsler-Krumeich classification The ICRS surgery was performed with the patient under topical anesthesia. A tunnel channel was created by femtosecond laser using a 60-kHz infrared neodymium glass femtosecond laser at a wavelength of 1053 nm (Abbott Laboratories Inc., Abbott Park, Illinois, USA). Two symmetrical kerarings (Mediphacos Inc., Belo Horizonte, Brazil), were implanted in all cases with 160° arc and 0.25, 0.30 mm according to corneal thickness in implantation site. After surgery, the patients had a full ocular evaluation on days 1, 7, and 14, and again after a month. For a period of 1-year, corneal topography readings were taken quarterly.

ELIGIBILITY:
Inclusion Criteria:

* stable keratoconus.
* corneal cross-linking performed at least 6 months.
* contact lens intolerance
* minimum corneal thickness of 350 μm at the thinnest point (TP)
* mean keratometry (K mean) value less than 59 D

Exclusion Criteria:

* any other associated ocular or systemic pathology could affect the vision.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
K1 and K2 post-operative by Pentacam | one year
  Flat and Steep K in Diopter post ring implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Elshimaa A.Mateen, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided